CLINICAL TRIAL: NCT04873219
Title: Evaluation of CAD/CAM Milled Versus Rapidly-prototyped (3D-printed) Complete Removable Dental Prostheses (CRDPs): a Double-blind Randomized Crossover Trial.
Brief Title: Milled Versus Printed CAD/CAM Complete Dentures
Acronym: MILLPRINT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Geneva, Switzerland (Other)
Responsible Party: Principal Investigator, Frauke Müller, Prof Dr med dent Dr hc Frauke Müller, University of Geneva, Switzerland
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: MDGPA_03
Record Dates: First submitted 2020-12-01; First posted 2021-05-05 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Denture, Complete; Jaw, Edentulous
Keywords: Computer-Aided Design; Computer-Assisted Manufacturing
MeSH Terms: conditions — Jaw, Edentulous

STUDY DESIGN:
Intervention Model Description: double blind single center cross-over design
Who Masked: Participant, Care Provider, Investigator
Masking Description: neither the patients, nor the operator knew which type of denture was inserted
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CAD/CAM milled complete denture (Active Comparator): the dentures were milled out of a block of pre-polymerized PMMA resin (Avadent, Global dental Science, Netherlands)
  Interventions: Device: manufacturing a complete dental prosthesis
- CAD/CAM rapid prototyped complete denture (Experimental): the dentures will be 3D-printed from a liquid PMMA, including the teeth (NexDent, Netherlands)
  Interventions: Device: manufacturing a complete dental prosthesis

INTERVENTIONS:
Device: manufacturing a complete dental prosthesis — dental treatment to replace missing teeth
  Other Names: complete denture manufacturing

SUMMARY:
A crossover clinical trial investigates two novel CAD/CAM techniques for complete removable dental prostheses for edentulous patients, milling and rapid prototyping (3D-printing) in a clinical setting of an undergraduate student clinic. Outcome parameters concern the dentures' trueness, retention, stability, esthetics and occlusion. Secondary outcome parameters include willingness to pay and prosthetic maintenance need.

DETAILED DESCRIPTION:
The process of fabricating complete removable dental prostheses (CRDPs) by novel CAD/CAM manufacturing technique has in the recent years gained immense popularity with clinicians as well as dental technicians worldwide. CRDPs can be manufactured by a subtractive process (milling technique) or by an additive process (rapid prototyping or 3D printing). The milling technique is the frequently employed technique for fabricating CRDPs; it is well documented in terms of precision, material properties, and a few clinical trials have even demonstrated good patient and clinician satisfaction. The rapid prototyping (3D printing) method however, is still in the developing stages for this particular application. Although both methods seem to yield clinically acceptable results, there are no studies in current literature which compare the CRDPs manufactured by the two CAD/CAM methods.

The proposed single-center, double-blind, randomized crossover clinical trial specifically aims to test the following hypothesis that:

• there is no difference between the two types of CRDPs (milled, and rapidly prototyped) in terms of trueness, denture quality, patient satisfaction, prosthodontic maintenance and adjustments requirements and incurred costs.

Fifteen pre-doctoral final year dental students and their respective completely edentulous patients will be recruited in this RCT. A traditional clinical complete denture protocol will be followed to record the clinical steps. Two sets of CRDPs will be manufactured (CAD/CAM milling and 3D printing). The CRDPs will be randomized before denture insertion and then delivered to the patient. Each CRDPs will be worn by the patient for a period of 6 weeks, before crossing over. Clinical examinations and data collection will be performed at baseline (T0), at denture insertion stage (T1), and at the end of 6 weeks (T2) for each of the investigated CRDPs. Assessments will comprise of comparison of trueness of denture intaglio surfaces against the corresponding master cast, denture quality assessments, patient satisfaction scores, prosthodontic maintenance needs and willingness-to-pay analysis and cost minimization analysis.

This RCT will contribute significantly in the development of CAD/CAM treatment concepts for fabricating complete removable dental prostheses (CRDPs). The study would highlight the differences, if any, between the two manufacturing methods for CRDPs, in terms of trueness, quality of the prostheses, clinician and patient satisfaction and also incurred costs. Clinically, the planned RCT hopes to demonstrate the feasibility of these novel treatment concepts in frail elderly edentates. A significant reduction in the treatment times, maintenance visits, and costs along with high patient satisfaction with these newer CRDPs would be added advantages when treating the elderly edentates.

ELIGIBILITY:
Inclusion Criteria:

* patient of undergraduate student at the University clinics of dental medicine Geneva
* completely edentulous
* requesting novel complete dentures

Exclusion Criteria:

* not willing to sign informed consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-09-15 (Actual); Primary Completion 2019-09-15 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Trueness of intaglio surface | Change from Baseline intaglio surface at 6-weeks
  fit of the dental prosthesis as evaluated by superimposition of scanned intaglio surfaces at baseline and at 6-weeks

SECONDARY OUTCOMES:
Clinician's denture quality | Change from Baseline denture retention and stability at 6-weeks
  denture quality questionnaire (Alfadda et al. 2014)
denture satisfaction Instrument | Change from Baseline denture satisfaction at 6-weeks
  patient's denture satisfaction questionnaire (Allen et al. 2001)
denture preference | after both dentures have been worn for 6 weeks
  the patient will decide which denture he/she prefers to keep after the clinical trial
prosthetic maintenance | at 6 weeks
  described adjustments and repair of the denture during the observation period
willingness to pay | at 6-weeks
  open ended contingency valuation method to evaluate the amount the patient would pay for the denture

CONTACTS AND LOCATIONS:
Overall Officials: Frauke Mueller, Prof Dr Dr, Principal Investigator — clinique universitaire de médecine dentaire
Locations (1):
- University clinics of dental medicine, Geneva, Canton of Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No